CLINICAL TRIAL: NCT05373485
Title: A Randomized, Double-blind, Dose-exploring, Placebo-controlled, Multi-center Phase I Clinical Trial Evaluating the Safety and Immunogenicity of COVID-19 mRNA Vaccine in Adults Aged 18 Years and Older
Brief Title: Phase I Clinical Trial of COVID-19 mRNA Vaccine in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-NCVM-001
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
Keywords: COVID; mRNA; Vaccine; Placebo; Safety; Immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Vaccine Group, low dose, 18-59 year-old (Experimental): 2 doses of COVID-19 mRNA vaccine (30µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Vaccine Group, low dose, 60 year-old and above (Experimental): 2 doses of COVID-19 mRNA vaccine (30µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Vaccine Group, high dose, 18-59 year-old (Experimental): 2 doses of COVID-19 mRNA vaccine (50µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Vaccine Group, high dose, 60 year-old and above (Experimental): 2 doses of COVID-19 mRNA vaccine (50µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: COVID-19 mRNA vaccine
- Placebo Group, low dose, 18-59 year-old (Placebo Comparator): 2 doses of placebo (0µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo
- Placebo Group, low dose, 60 year-old and above (Placebo Comparator): 2 doses of placebo (0µg, 0.3 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo
- Placebo Group, high dose, 18-59 year-old (Placebo Comparator): 2 doses of placebo (0µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo
- Placebo Group, high dose, 60 year-old and above (Placebo Comparator): 2 doses of placebo (0µg, 0.5 ml) on Day 0 and Day 21
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: COVID-19 mRNA vaccine — 2 doses of vaccine on Day 0 and Day 21
  Arms: Vaccine Group, high dose, 18-59 year-old; Vaccine Group, high dose, 60 year-old and above; Vaccine Group, low dose, 18-59 year-old; Vaccine Group, low dose, 60 year-old and above
Biological: Placebo — 2 doses of placebo on Day 0 and Day 21
  Arms: Placebo Group, high dose, 18-59 year-old; Placebo Group, high dose, 60 year-old and above; Placebo Group, low dose, 18-59 year-old; Placebo Group, low dose, 60 year-old and above

SUMMARY:
To evaluate the safety and immunogenicity of the COVID-19 mRNA vaccine in people aged 18 years and older, 80 participants will be enrolled and divided into two groups: low- and high-dose groups. Each dose group will be divided into 2 age groups (20 people each):18 to 59 years old and ≥ 60 years old. Subjects will be randomized into vaccine group or placebo group in a ratio of 3:1. Subjects will receive 2 doses of either vaccine or placebo on Day 0 and Day 21, in which the low-dose group will received 0.3 ml of the study vaccine or placebo, and the high dose group will receive 0.5 ml of the study vaccine or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above with BMI of 18 to 30 (including boundary values);
2. Volunteers are able and willing to comply with the requirements of the clinical trial protocol, and volunteers or witnesses can sign informed consent forms;
3. Willing to discuss the medical history with the investigator or doctor and allow access to all medical records related to this trial;
4. Provide 48-hour PCR negative report;
5. Have not received any other COVID-19 vaccines.

Exclusion Criteria:

* Criteria for exclusion of the first dose

  1. Other medical or psychiatric conditions, including recent (within the past year) or current presence of suicidal ideation/behavior, or laboratory abnormalities that may increase the risk of participating in the study, or subjects who are not suitable to participate in the study according to the investigator's judgment;
  2. Positive for human immunodeficiency virus (HIV);
  3. History of infection or disease of Middle East Respiratory Syndrome (MERS), SARS or other coronaviruses or related immunizations;
  4. History of serious adverse reactions associated with the vaccine and/or a history of severe allergic reactions (e.g., anaphylaxis) to any component of the vaccine under study;
  5. Immunocompromised patients with known or suspected immunodeficiency identified by medical history and/or physical examination;
  6. Bleeding constitution or condition associated with prolonged bleeding which investigators believe that intramuscular injection is contraindicated;
  7. Women who test positive for blood pregnancy or are breastfeeding, volunteers or their partners have a pregnancy plan within 12 months;
  8. Severe hypertension and uncontrollable medication (on-site measurement: systolic blood pressure ≥ 160mmHg, diastolic blood pressure ≥ 100mmHg);
  9. Have a serious chronic disease or the condition is in the progression period can not be smoothly controlled, such as diabetes, thyroid disease, etc.;
  10. History of severe myocarditis, pericarditis and other heart diseases;
  11. Abnormal laboratory tests during the screening window and judged by researchers to be of clinical significance;
  12. Plans to receive other vaccines within 28 days before and after receiving the test vaccine;
  13. Those receiving immunosuppressive therapy, including cytotoxic drugs or systemic corticosteroids, such as for cancer or autoimmune diseases, or who were scheduled to receive treatment throughout the study period. If systemic corticosteroids are used in a short period of time (< 14 days) for the treatment of acute illness, subjects should not enter this study until at least 28 days after corticosteroid therapy has been discontinued prior to study vaccination. Inhalation/spraying, intra-articular, intraskeletal, or topical (skin or eyes) use of corticosteroids is permitted;
  14. Receiving blood/plasma products or immunoglobulins 60 days prior to study vaccination or plan to receive for the entire study duration;
  15. Engage in other interventional studies within 28 days prior to entering the study and/or during the study's participation;
  16. Participated in other interventional studies of lipid-containing nanoparticles;
  17. Have symptoms of COVID-19 such as respiratory symptoms, fever, cough, shortness of breath, and dyspnea;
  18. Fever, axillary temperature > 37.0 °C.

Second dose exclusion criteria:

1. Severe allergic reactions occur after the first vaccination;
2. Serious adverse reactions with causal relationship during the first vaccination;
3. Those who are newly discovered or newly occurring after the first vaccination do not meet the inclusion criteria of the first dose or meet the exclusion criteria of the first dose, and the investigator shall decide whether to continue to participate in the study;
4. Other reasons for exclusion that the investigators believe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse reactions (AR) | within 14 days of immunization
  To evaluate the incidence of adverse reactions (AR) within 14 days of immunization in all subjects

SECONDARY OUTCOMES:
The incidence of adverse reactions (AR) | within 28 days of immunization
  To evaluate the incidence of adverse reactions (AR) within 28 days of immunization in all subjects
The incidence of SAE, MAE and AESI | From vaccination to post of 12 months vaccination
  To evaluation the incidence of SAE, MAE, and AESI within 12 months of full immunization in all subjects
The incidence of adverse reactions (AR) | Within 60 minutes of each vaccination
  To evaluate the incidence of adverse reactions (AR) within 60 minutes of each vaccination in all subjects
Changes in laboratory indicators | Day 4 and Day 7 post each vaccination
  Changes in white blood cell count
Changes in laboratory indicators | Day 4 and Day 7 post each vaccination
  Changes in neutrophils
Changes in laboratory indicators | Day 4 and Day 7 post each vaccination
  Changes in lymphocyte count;
Changes in laboratory indicators | Day 4 and Day 7 post each vaccination
  Changes in platelet count;
Immunogenicity of wild type neutralizing antibodies | Before the 2nd dose, 14 days after the 2nd dose, and 28 days after the 2nd dose
  Sero-conversation rate of anti-wild type neutralizing antibodies
Immunogenicity of wild type neutralizing antibodies | Before the 2nd dose, 14 days after the 2nd dose, and 28 days after the 2nd dose
  Geometric mean titer (GMT) of wild type neutralizing antibodies
Immunogenicity of wild type neutralizing antibodies | Before the 2nd dose, 14 days after the 2nd dose, and 28 days after the 2nd dose
  GMI of wild type neutralizing antibodies
Immunogenicity of anti-S-RBD Ig G antibodies | Before the 2nd dose, 14 days after the 2nd dose, and 28 days after the 2nd dose
  Sero-conversation rate of anti-S-RBD Ig G antibodies
Immunogenicity of anti-S-RBD Ig G antibodies | Before the 2nd dose, 14 days after the 2nd dose, and 28 days after the 2nd dose
  GMC of anti-S-RBD Ig G antibodies
Immunogenicity of anti-S-RBD Ig G antibodies | Before the 2nd dose, 14 days after the 2nd dose, and 28 days after the 2nd dose
  GMI of anti-S-RBD Ig G antibodies
Changes in vital signs | Day 1 to 4 , Day 7 after the first dose, and the day of second dose, Day 4 after the second dose, and day 7 after the second dose
  The incidence of outliers detected on vital signs
Immuno-persistency of wild type neutralizing antibodies | Month 3,6 and 12 post second vaccination
  Sero-conversation rate of anti-wild type virus neutralizing antibodies
Immuno-persistency of wild type neutralizing antibodies | Month 3,6 and 12 post second vaccination
  GMT of wild type neutralizing antibodies
Immuno-persistency of wild type neutralizing antibodies | Month 3,6 and 12 post second vaccination
  GMI of wild type neutralizing antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Dong, Principal Investigator — Beijing Friendship Hospital; Kexin Zhao, Principal Investigator — Hebei Petro China Center Hospital; Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Hebei Petro China Center Hospital, Langfang, Hebei
  - Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan

REFERENCES:
- [Derived] Jin Z, Wu J, Wang Y, Huang T, Zhao K, Liu J, Wang H, Zhu T, Gou J, Huang H, Wu X, Yin H, Song J, Li R, Zhang J, Li L, Chen J, Li X, Zhang M, Li J, Hou M, Song Y, Wang B, Gao Q, Wu L, Kong Y, Dong R. Safety and immunogenicity of the COVID-19 mRNA vaccine CS-2034: A randomized, double-blind, dose-exploration, placebo-controlled multicenter Phase I clinical trial in healthy Chinese adults. J Infect. 2023 Dec;87(6):556-570. doi: 10.1016/j.jinf.2023.10.012. Epub 2023 Oct 28. PMID 37898410